## Assessing the Feasibility of Economic Approaches to Prevent Substance Abuse Among Adolescents

NCT Number: NCT05597865

Statistical analysis plan updated June 20th 2025

The primary study outcomes were feasibility and acceptability of the research protocol, assessed using a mixed methods approach. Quantitatively, feasibility will be determined by the proportion of participants who enrolled in the intervention. Acceptability will be determined by measuring retention rates at 6 months, adherence to study procedures, intervention attendance and engagement. To assess whether participants adhered to and engaged in the intervention components we will report descriptive statistics to track the number and percentage of participants completing each intervention session, and the retention rate at the 6-month follow-up.

To examine short-term outcomes of the randomized controlled trial (RCT), with a focus on changes in prevalence of alcohol and drug use and psychosocial variables from baseline to 6-months. Categorical variables will be summarized using counts and percentages, and continuous outcomes will be summarized using means and standard deviation (SD) for the overall group and by study arm. Following noted experts and NIH guidance, we acknowledge that pilot RCT studies are too small to allow for sufficiently powered statistical tests or reliable effect size estimates to be determined or to conduct formal tests of clinical outcomes. In addition, attempting to obtain precise estimates of effect sizes cannot be statistically justified. Thus, in this pilot RCT we will focus on feasibility and acceptability of the protocol- design and adjustments necessary to maximize recruitment, retention, and quality assessment of outcomes in future studies.